CLINICAL TRIAL: NCT04241523
Title: Efficacy and Safety of Lenvatinib as a Conversion Therapy in Patients With Potentially Resectable Hepatocellular Carcinoma: A Single-Arm and Open-Label Prospective Study
Brief Title: Efficacy and Safety of Lenvatinib as a Conversion Therapy for HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Tongji Hospital (Other); Anhui Provincial Hospital (Other Government); West China Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Professor of Surgery, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-LEN-Conversion
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): The patients will receive lenvatinib treatment and will be evaluated for the feasibility of liver resection every 8 weeks. For those who underwent liver resection, they will receive lenvatinib treatment for another 48 weeks. In case of tumor recurrence, intolerance, death, or need for other antitumor treatment, the treatment shall be stopped.
  Interventions: Drug: Lenvatinib 4 mg Oral

INTERVENTIONS:
Drug: Lenvatinib 4 mg Oral — Planned doses of 8 mg of lenvatinib per day for patients with body weight <60 kg, and 12 mg for those with body weight ≥60 kg.
  In case of treatment-related adverse effects, interruption or reduction is allowed.
  Other Names: Lenvima 4 mg Oral

SUMMARY:
Lenvatinib is the standard of care for patients with advanced hepatocellular carcinoma (HCC). The aim of the single-arm, open-label, phase II clinical trial is to assess efficacy and safety of lenvatinib as a preoperative conversion therapy in patients with potentially resectable HCC. Investigator hypothesized that lenvatinib may be an effective conversion treatment for HCC, and preoperative treatment with lenvatinib can improve resectability in patients with potential resectable HCC and improve the long term survival.

DETAILED DESCRIPTION:
For patients with potentially resectable HCC (intermediate or advanced stage), upfront therapy with surgical resection is of high recurrence rate after surgery. The aim of the single-arm, open-label, prospective phase II clinical trial is to evaluate whether preoperative lenvatinib treatment could improve resectability and therefore improve the long term survival.

Participants who are recruited in this study in this study will be treated with lenvatinib and will be evaluated for the feasibility for surgical resection by a multidisciplinary team every 8 weeks. If the participants underwent curative resection, they will receive lenvatinib treatment for 48 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75;
2. The participant must have confirmed diagnosis of HCC histologically or clinically;
3. The participant must have at least one untreated intrahepatic lesion that can be evaluated by contrast-enhanced CT or MRI;
4. The BCLC stage B/C patients, more than 3 tumor nodes or have portal vein tumor thrombus (Vp3-Vp4 according to LCSGJ PVTT classification) or extrahepatic metastases limited to one organ and the number of metastases nodules is no more than 3;
5. ECOG PS 0-1 and Child-Pugh A;
6. Surgical resection is not the first choice according to MDT evaluation;
7. Written informed consent;

Exclusion Criteria:

1. WBC<4.0*10^9/L, HB<80 g/L, PLT<75*10^9/L and NEUT<1.5×10^9/L;
2. Coagulation function: (prothrombin time) international normalized ratio (INR) >1.2;
3. Liver function: serum albumin (ALB)<3.5 g/dl, total bilirubin (TBIL)>1.5 times the upper limit of normal range, alanine aminotransferase and aspartate aminotransferase (ALT and AST)>3 times the upper limit of normal range; renal function index: serum creatinine (CRE)>1.5 times the upper limit of normal range; uncontrolled hypertension (>150/90mm Hg);
4. Lymph node metastasis to hilar of lung or liver, or peripheral tissue adhesion;
5. Participated in other clinical trials 30 days before enrollment;
6. With ascites, hepatic encephalopathy, Gilbert syndrome, sclerosing cholangitis;
7. Suspected allergy to study drug;
8. With other organ dysfunction, it is not expected to be tolerated general anesthesia or hepatectomy;
9. Other conditions that the investigators considered not unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Resection rate | 1 year after LPI
  The percentage of patients who receive curative liver resection for HCC. The criteria for curative resection: (1) no active tumor thrombosis is observed in hepatic veins, portal veins, bile ducts or inferior vena cava; or the type of portal vein invasion was converted from Vp3/Vp4 to Vp1/Vp2; (2) no active metastasis to adjacent organs or distant organs, or to lymph nodes; (3) the surgical margin ≥ 0.5 cm; (4) the number of active tumor nodules decreases from ≥4 to <4; (5) the ratio of future liver volume to standard liver volume increases from <40% to ≥40% (for those with liver cirrhosis) or from <30% to ≥30% (for those without liver cirrhosis).

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  The duration from the date of recruitment to the date of death from any cause.
Objective response rate (ORR) | 1 year after LPI
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters)
Serum Biomarkers | 1 year after LPI
  To explore the relationship between the baseline level and dynamic changes of serum markers(AFP and PIVKA-II) and therapeutic response, Peripheral blood serum was collected at baseline and at each follow-up visit.
Adverse events(AE) and Serious adverse events(SAE) | 1 year after LPI
  An adverse event (AE) refers to any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, but which does not necessarily have a causal relationship with this treatment.
  A serious adverse event (SAE) refers to an event in clinical trials that requires inpatient hospitalization or causes prolongation of existing hospitalization, permanent disability, incapacity, threats to life or death, and birth defect, etc.
  Number and classification of participants with treatment-related adverse events as assessed by CTCAE v4.0 were recorded.
Health-related quality of life: EORTC QLQ-HCC18 | 1 year after LPI
  Health-related quality of life questionnaire measured by EORTC QLQ-HCC18.
Exploratory serum biomarker research | 1 year after LPI
  About 10 mL peripheral blood will be collected at baseline and at each follow-up visit. The correlations between serum biomarkers at baseline or the dynamic changes and treatment response will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Principal Investigator — Shanghai Zhongshan Hospital
Locations (4):
- China (4):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Tongji Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - West China Hospital, Chengdu, Sichuan
  - 180 Fenglin Road, Shanghai

IPD SHARING:
Plan to Share IPD: No